CLINICAL TRIAL: NCT03166709
Title: Preventing Addiction Related Suicide (PARS) - Controlled Trial of Secondary Suicide Prevention
Brief Title: Preventing Addiction Related Suicide (PARS)
Acronym: PARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kate Comtois, Professor, Dept of Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001966; 1R01DA041486-01A1 (NIH)
Record Dates: First submitted 2017-05-22; First posted 2017-05-25 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Suicide; Substance-Related Disorders
MeSH Terms: conditions — Suicide; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Stepped wedge - 15 sites randomly divided into 5 groups which are then randomly ordered into 5 steps. Step 1 is all control. During steps 2-6 one group implements the experimental condition in assigned order until all groups are doing experimental condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (Active Comparator): Intensive Outpatient Program (IOP) addiction treatment
  Interventions: Behavioral: Intensive Outpatient Program standard session
- Experimental (Experimental): Secondary Prevention Intervention (PARS) plus Treatment as Usual
  Interventions: Behavioral: Preventing Addiction Related Suicide (PARS)

INTERVENTIONS:
Behavioral: Preventing Addiction Related Suicide (PARS) — PARS is a module designed for a single session of an Intensive Outpatient Program (IOP) including a specified combination of didactic presentations and group discussions. PARS topics include: Goals and Objectives; Suicide Overview; The Strong Link Between Addiction and Suicide; Suicide Myths and Facts; Common Triggers of Suicidal Thoughts and Behaviors; Warning Signs of Suicide; Suicide Risk Factors; Suicide Protective Factors; How You Can Prevent Addiction Related Suicide; Action Steps to Take if You or Someone You Know Becomes Suicidal
  Arms: Experimental
Behavioral: Intensive Outpatient Program standard session — Intensive Outpatient Program (IOP) substance abuse group session focused on depression, grief, or managing emotions. Site-specific session topic is what that IOP usually provides and was chosen by agency leads prior to start of study.
  Arms: Treatment As Usual

SUMMARY:
The goal of this study is to evaluate the effectiveness and utility of the investigator's National Institute on Drug Abuse (NIDA) R21 developed "Preventing Addiction Related Suicide" (PARS) program by utilizing a novel stepped wedge design to evaluate PARS as a selected prevention program to increase help-seeking by clients in community addiction treatment.

DETAILED DESCRIPTION:
Studies consistently show suicide and suicidal behaviors are highly related to substance use disorders (SUDs). Recent reviews find that the risk of suicide is 10-17 times higher for people using multiple drugs, injecting drugs, and for alcohol use disorders. SUDs are also related to suicidal thoughts and suicide attempts. Clients admitted for alcohol treatment report a much higher rate of lifetime suicide attempts (40-43%) than a nationally representative sample of adults (4.6%). Further, prospective data shows that individuals in addiction treatment had five times the odds of suicide attempt over five years compared to those not in treatment, emphasizing addiction treatment as a key opportunity for instituting suicide prevention strategies.

Based on Stage I guidelines for developing and adapting behavioral interventions and information from a Substance Abuse and Mental Health Services Administration (SAMHSA) Treatment Improvement Protocol (TIP50) on suicide and addiction, we developed the Preventing Addiction Related Suicide (PARS) program.

To maximize the chances of implementation, PARS was developed to be a community-friendly program with a team of community partners (i.e., administrators, counselors, clients) who advised on its scope, duration, and approach. Community leaders reviewed PARS throughout its development and pilot testing was conducted in their community treatment settings. Thus, PARS is simultaneously based on evidence-based practice and the goals and needs of community treatment settings. Importantly, PARS is a selected prevention program and not intervention for suicidality per se-it is designed for all clients in addiction treatment as a standard part of care. PARS' goal is increased help-seeking by addiction treatment clients as well as by clients' friends and family if and when they themselves become suicidal. Reaching out for help leads to care that can address and resolve suicidality. PARS is the only published selected prevention program for this high-risk population.

PARS is a psychoeducational program taught as a single three-hour module integrated into a standard group therapy-oriented Intensive Outpatient Program (IOP), the most common form of community addiction treatment. Pilot testing of PARS in three community agencies demonstrated significant post-intervention increases in accurate information about suicide and decreases in maladaptive attitudes toward suicide. These changes at post-intervention were maintained at 1-month follow-up. Even more compelling, 1-month follow-up assessments demonstrated that the likelihood of positive help seeking for suicidality doubled for the month after PARS compared to the month before. Clients were significantly more likely to ask suicidal friends (from 9% to 22%) and family (9% to 17%) to seek help as well as to seek help themselves (4% to 9%).

Given these promising Stage I results in Stage III settings, we propose a fully-powered Stage III effectiveness trial of PARS compared to Treatment-as-Usual (TAU) using a stepped wedge design with 900 clients enrolled in 15 community addiction treatment sites. We will collect outcome data post-intervention and at 1, 3, and 6 months follow-up. We propose the following research aims:

Aim 1: Compare the effectiveness of IOP integrating PARS to TAU to change beliefs about suicide and suicide prevention.

Hypothesis 1a: Clients who receive PARS will know more accurate information about suicide.

Hypothesis 1b: Clients who receive PARS will have less maladaptive attitudes about suicide.

Aim 2: Compare the effectiveness of IOP integrating PARS to TAU to increase help-seeking behaviors for clients and for clients' friends or family at risk of suicide.

Hypothesis 1c: Clients who receive PARS will show greater help-seeking for themselves and others

Aim 3: Evaluate whether changes in beliefs about suicide and suicide prevention-particularly regarding warning signs for suicide, including addiction, intoxication, and relapse, as well as beliefs that suicide is preventable when action is taken-are possible mechanisms by which PARS increases help-seeking behavior.

Hypothesis 2: The effect of PARS vs. TAU on changes in help-seeking will be mediated by improved information and attitudes.

Exploratory Aim 4: Evaluate possible clinic-level dose effects of PARS administration such that participant outcomes improve the longer PARS is implemented within clinics.

Exploratory Aim 5: Compare the effects of PARS vs. TAU on clients' suicidality and substance use in the follow-up period.

By integrating PARS into IOP group treatment, community treatment agencies are in a unique position to act as key players in the national suicide prevention strategy by providing suicide prevention information, improving attitudes regarding suicide, and increasing help-seeking skills for one of the most high-risk populations for suicide. This proposal is innovative in its focus, the development of PARS in community settings, as well as the use of a stepped wedge design.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled client in one of the community treatment settings
2. Over 18 years of age (no maximum age)
3. Ability to understand written and spoken English

Exclusion Criteria:

1. Any clinical medical/psychiatric condition, severity of that condition, or life situation that in the opinion of the counselors or Drs. Comtois or Ries would compromise safe and voluntary study participation (e.g., psychosis, custody conflict). This is expected to be a rare circumstance and will be known prior to the recruitment session. If a counselor does not want someone involved, they will not be. If counselor is unsure, Dr. Comtois or Ries will facilitate decision with counselor ahead of time to assist in the decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Anne Comtois, PhD, MPH, Principal Investigator — University of Washington
Locations (16):
- United States (16):
  - Lakeside-Milam, Auburn, Washington
  - Lakeside-Milam, Edmonds, Washington
  - Evergreen Recovery Centers, Everett, Washington
  - Lakeside-Milam, Everett, Washington
  - Olalla Recovery Centers, Gig Harbor, Washington
  - Lakeside-Milam, Issaquah, Washington
  - Lakeside-Milam, Kirkland, Washington
  - Northwest Integrated Health, Lakewood, Washington
  - Evergreen Recovery Centers, Lynnwood, Washington
  - Lakeside-Milam, Puyallup, Washington
  - Northwest Integrated Health, Puyallup, Washington
  - Lakeside-Milam, Renton, Washington
  - Lakeside-Milam, Seattle, Washington
  - THS, Seattle, Washington
  - Lakeside-Milam, Tacoma, Washington
  - Northwest Integrated Health, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ries RK, Livengood AL, Huh D, Kerbrat AH, Fruhbauerova M, Turner B, Comtois KA. Effectiveness of a Suicide Prevention Module for Adults in Substance Use Disorder Treatment: A Stepped-Wedge Cluster-Randomized Clinical Trial. JAMA Netw Open. 2022 Apr 1;5(4):e222945. doi: 10.1001/jamanetworkopen.2022.2945. PMID 35385090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment completed between October 2017 and September 2019
Units Other Than Participants: Site
Groups:
- Group 1: 4 Months TAU, 20 Months PARS: Group 1: 90 day Intensive Outpatient Program - 4 months Treatment as Usual (Control Condition), 20 months PARS (Experimental Condition).
- Group 2: 8 Months TAU, Then 16 Months PARS: Group 2: 90 day Intensive Outpatient Program - 8 months Treatment as Usual (Control Condition), 16 months PARS (Experimental Condition)
- Group 3: 12 Months TAU,12months PARS: Group 3: 90 day Intensive Outpatient Program - 12 months Treatment as Usual (Control Condition), 12 months PARS (Experimental Condition)
- Group 4: 16 Months TAU, 8 Months PARS: Group 4: 90 day Intensive Outpatient Program - 8 months Treatment as Usual (Control Condition), 16 months PARS (Experimental Condition)
- Group 5: 20 Months TAU, 4 Months PARS: Group 5: 90 day Intensive Outpatient Program - 20 months Treatment as Usual (Control Condition), 4 months PARS (Experimental Condition)
Period: Step 1 (Months 1-4)
Arm/Group | Group 1: 4 Months TAU, 20 Months PARS | Group 2: 8 Months TAU, Then 16 Months PARS | Group 3: 12 Months TAU,12months PARS | Group 4: 16 Months TAU, 8 Months PARS | Group 5: 20 Months TAU, 4 Months PARS
Started | 29; 3 Site | 38; 3 Site | 39; 3 Site | 42; 3 Site | 38; 3 Site
Completed | 23; 3 Site | 24; 3 Site | 23; 3 Site | 25; 3 Site | 27; 3 Site
Not Completed | 6; 0 Site | 14; 0 Site | 16; 0 Site | 17; 0 Site | 11; 0 Site
Period: Step 2 (Months 5-8)
Arm/Group | Group 1: 4 Months TAU, 20 Months PARS | Group 2: 8 Months TAU, Then 16 Months PARS | Group 3: 12 Months TAU,12months PARS | Group 4: 16 Months TAU, 8 Months PARS | Group 5: 20 Months TAU, 4 Months PARS
Started | 23; 3 Site (New participants were recruited in each period (aka step).) | 34; 3 Site (New participants were recruited in each period (aka step).) | 21; 3 Site (New participants were recruited in each period (aka step).) | 37; 3 Site (New participants were recruited in each period (aka step).) | 34; 3 Site (New participants were recruited in each period (aka step).)
Completed | 19; 3 Site | 28; 3 Site | 16; 3 Site | 23; 3 Site | 25; 3 Site
Not Completed | 4; 0 Site | 6; 0 Site | 5; 0 Site | 14; 0 Site | 9; 0 Site
Period: Step 3 (Months 9-12)
Arm/Group | Group 1: 4 Months TAU, 20 Months PARS | Group 2: 8 Months TAU, Then 16 Months PARS | Group 3: 12 Months TAU,12months PARS | Group 4: 16 Months TAU, 8 Months PARS | Group 5: 20 Months TAU, 4 Months PARS
Started | 23; 3 Site (New participants were recruited in each period (aka step).) | 28; 3 Site (New participants were recruited in each period (aka step).) | 26; 3 Site (New participants were recruited in each period (aka step).) | 27; 3 Site (New participants were recruited in each period (aka step).) | 24; 3 Site (New participants were recruited in each period (aka step).)
Completed | 19; 3 Site | 17; 3 Site | 19; 3 Site | 12; 3 Site | 18; 3 Site
Not Completed | 4; 0 Site | 11; 0 Site | 7; 0 Site | 15; 0 Site | 6; 0 Site
Period: Step 4 (Months 13-16)
Arm/Group | Group 1: 4 Months TAU, 20 Months PARS | Group 2: 8 Months TAU, Then 16 Months PARS | Group 3: 12 Months TAU,12months PARS | Group 4: 16 Months TAU, 8 Months PARS | Group 5: 20 Months TAU, 4 Months PARS
Started | 27; 3 Site (New participants were recruited in each period (aka step).) | 29; 3 Site (New participants were recruited in each period (aka step).) | 26; 3 Site (New participants were recruited in each period (aka step).) | 26; 3 Site (New participants were recruited in each period (aka step).) | 34; 3 Site (New participants were recruited in each period (aka step).)
Completed | 22; 3 Site | 23; 3 Site | 17; 3 Site | 13; 3 Site | 26; 3 Site
Not Completed | 5; 0 Site | 6; 0 Site | 9; 0 Site | 13; 0 Site | 8; 0 Site
Period: Step 5 (Months 17-20)
Arm/Group | Group 1: 4 Months TAU, 20 Months PARS | Group 2: 8 Months TAU, Then 16 Months PARS | Group 3: 12 Months TAU,12months PARS | Group 4: 16 Months TAU, 8 Months PARS | Group 5: 20 Months TAU, 4 Months PARS
Started | 34; 3 Site (New participants were recruited in each period (aka step).) | 32; 3 Site (New participants were recruited in each period (aka step).) | 31; 3 Site (New participants were recruited in each period (aka step).) | 29; 3 Site (New participants were recruited in each period (aka step).) | 29; 3 Site (New participants were recruited in each period (aka step).)
Completed | 25; 3 Site | 21; 3 Site | 24; 3 Site | 17; 3 Site | 21; 3 Site
Not Completed | 9; 0 Site | 11; 0 Site | 7; 0 Site | 12; 0 Site | 8; 0 Site
Period: Step 6 (Months 21-24)
Arm/Group | Group 1: 4 Months TAU, 20 Months PARS | Group 2: 8 Months TAU, Then 16 Months PARS | Group 3: 12 Months TAU,12months PARS | Group 4: 16 Months TAU, 8 Months PARS | Group 5: 20 Months TAU, 4 Months PARS
Started | 41; 3 Site (New participants were recruited in each period (aka step).) | 27; 3 Site (New participants were recruited in each period (aka step).) | 25; 3 Site (New participants were recruited in each period (aka step).) | 22; 3 Site (New participants were recruited in each period (aka step).) | 31; 3 Site (New participants were recruited in each period (aka step).)
Completed | 27; 3 Site | 13; 3 Site | 18; 3 Site | 11; 3 Site | 20; 3 Site
Not Completed | 14; 0 Site | 14; 0 Site | 7; 0 Site | 11; 0 Site | 11; 0 Site

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment As Usual | Experimental | Total
Number analyzed (Participants) | 478 | 428 | 906
Age, Categorical [Count of Participants; unit: Participants] — Population: 40 participants did not provide their age
  Participants
    number analyzed (Participants) | 450 | 416 | 866
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 445 | 411 | 856
    >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 40 participants did not provide their age
  years
    number analyzed (Participants) | 450 | 416 | 866
    (all) | 37.3 (12.4) | 37.7 (11.7) | 37.5 (12.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Women | 201 | 149 | 350
  Men | 269 | 271 | 540
  Transexual or Non-Conforming Transgender or nonconforming | 2 | 2 | 4
  Unknown | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 42 | 73
  Not Hispanic or Latino | 439 | 378 | 817
  Unknown or Not Reported | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 10 | 26
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 6 | 2 | 8
  Black or African American | 16 | 17 | 33
  White | 347 | 326 | 673
  More than one race | 62 | 46 | 108
  Unknown or Not Reported | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  United States | 478 | 428 | 906
PARS Suicide Knowledge Scale [Mean (Standard Deviation); unit: units on a scale] — The PARS Suicide Knowledge Scale is an 11-item measure adapted from the Staff Suicide Prevention Survey (SSPS) assessing factual understanding of suicide and closely mapped to the content of PARS. Correct responses were summed to create a score from 0 to 11. Previous research demonstrated validity pre- and post-suicide training and test-retest reliability from baseline to post-treatment in the TAU condition ranged from 0.46-0.62.
  units on a scale | 7.42 (1.68) | 7.76 (1.70) | 7.58 (1.69)
PARS Attitude Scale [Mean (Standard Deviation); unit: units on a scale] — The PARS Attitude Scale, also adapted from the Staff Suicide Prevention Survey (SSPS), consists of 6 items evaluating attitudes about suicide stigma and prevention. Responses on a 5-point scale from "strongly disagree" (=1) to "strongly agree" (=5) were summed to create a score from 6 to 30. Internal consistency based on the pilot sample was 0.73-0.97 and in this full sample was 0.59-0.73.
  units on a scale | 12.81 (3.25) | 12.58 (3.38) | 12.70 (3.32)
PARS Help-Seeking Scale [Mean (Standard Deviation); unit: units on a scale] — The PARS Help-Seeking Scale consists of 4 items assessing help-seeking behavior in the context of suicidal thoughts or feelings (e.g., calling a crisis/suicide hotline) developed for our pilot trial based on prior suicide prevention programs. Participants reported the frequency of past-month help-seeking on behalf of self or others, including friends and family members, from "never" (=0) to "more than 3 times" (=4). Responses were summed to create a score from 0 to 16. Internal consistency based on the pilot sample was 0.82-0.87 and in this full sample was 0.52-0.76.
  units on a scale | 0.63 (1.45) | 0.48 (1.14) | 0.56 (1.32)

OUTCOME MEASURES:

1. Primary Outcome: PARS Help-Seeking Scale
Description: The PARS Help-Seeking Scale consists of 4 items assessing help-seeking behavior in the context of suicidal thoughts or feelings (e.g., calling a crisis/suicide hotline) developed for our pilot trial22 based on prior suicide prevention programs. Participants reported the frequency of past-month help-seeking on behalf of self or others, including friends and family members, from "never" (=0) to "more than 3 times" (=4). Responses were summed to create a score from 0 to 16 with higher numbers indicating the better outcome of increased help-seeking.
Time Frame: Six months
Population: Missing data for 107 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment As Usual | Experimental
Number analyzed (Participants) | 411 | 388
units on a scale | 0.57 (1.54) | 0.53 (1.66)

2. Primary Outcome: PARS Suicide Knowledge Scale
Description: The PARS Suicide Knowledge Scale is an 11-item measure adapted from the Staff Suicide Prevention Survey (SSPS) assessing factual understanding of suicide and closely mapped to the content of PARS. Correct responses were summed to create a score from 0 to 11 with higher scores representing the better outcome of greater suicide knowledge.
Time Frame: Six months
Population: Missing data from 95 participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment As Usual | Experimental
Number analyzed (Participants) | 420 | 391
units on a scale | 7.47 (1.89) | 8.24 (1.83)

3. Primary Outcome: PARS Attitude Scale
Description: The PARS Attitude Scale, adapted from the Staff Suicide Prevention Survey (SSPS), consists of 6 items evaluating maladaptive attitudes about suicide stigma and prevention. Responses on a 5-point scale from "strongly disagree" (=1) to "strongly agree" (=5) were summed to create a score from 6 to 30 where lower scores indicate a better outcome.
Time Frame: Six months
Population: Missing data for 121 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment As Usual | Experimental
Number analyzed (Participants) | 403 | 382
units on a scale | 12.29 (3.60) | 11.14 (3.88)

4. Secondary Outcome: Suicidal Behavior Questionnaire - Revised
Description: The Suicidal Behavior Questionnaire - Revised assesses suicide attempts, ideation, communication, and intent since the last assessment. Total score with higher indicating the worse outcome of suicide risk from lowest (3) to highest (18); non-clinical cutoff 7 and above
Time Frame: Six months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment As Usual | Experimental
Number analyzed (Participants) | 478 | 428
units on a scale | 4.54 (2.19) | 4.82 (2.41)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment As Usual | Experimental
All-Cause Mortality (participants affected / at risk) | 4/478 | 1/428
Serious Adverse Events (participants affected / at risk) | 4/478 | 1/428
Other Adverse Events (participants affected / at risk) | 0/478 | 0/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment As Usual (N=478) | Experimental (N=428)
Suicide Attempt, Psychiatric Hospitalization or Any Death (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) — NIH definition of SAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03166709/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03166709/SAP_001.pdf